CLINICAL TRIAL: NCT04209413
Title: Control of the Opening of mPTP by Ex Vivo Measurements on Permeabilized Muscle Fibers
Brief Title: Control of the Opening of mPTP by Ex Vivo Measurements on Permeabilized Muscle Fibers (COMMEF)
Acronym: COMMEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government)
Responsible Party: Sponsor
Other Study IDs: RNI 2019 RICHARD; 2019-A01109-48 (Other: ANSM)
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Anterior Cruciate Ligament operation; Skeletal muscle; Mitochondria; Calcium; Mitochondrial permeability transition pore opening (mPTP opening)
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Patients referred for a knee ligamentoplasty — knee ligamentoplasty

SUMMARY:
mPTP (Mitochondrial Permeability Transition Pore) is a channel formed by a protein complex integrated into the inner membrane of mitochondria. Its opening is related to the elevation of the intra-mitochondrial calcium concentration and will result in: a mitochondrial decoupling, a rupture of the metabolic gradient and the release of pro-apoptotic factors.

The objective of this study is the development of a new ex vivo technique for characterizing mPTP by a dual measurement combining oxygraphy and fluorimetry on permeabilized skeletal muscle fibers.

DETAILED DESCRIPTION:
The development of new expertise in the study of mPTP is part of an approach to optimize the processing of muscle samples. The aim of this work is to evaluate the feasibility and reproducibility of a method of analysis on muscle fibers only permeabilized, while coupling two complementary techniques, oxygraphy and fluorimetry. Its principle is based on the knowledge that the opening of the mPTP leads to an inhibition of respiration at the level of the complex I of the respiratory chain. This inhibition is the consequence of the escape from mitochondria of the reduced form of nicotinamide adenine dinucleotide (NADH, i.e. substrate of complex I) concomitant with the opening of mPTP. Thus, the oxygraphy must allow the observation of the inhibition of respiration synonymous with the non-availability of the substrate of the complex I and thus indirectly reflect the opening of the mPTP. For its part, the fluorimetry must allow, in the presence of a fluorescent calcium indicator (i.e. Calcium Green), the observation of the release of calcium synonymous with the opening of the mPTP.

Once validated, this technique should make it possible to evaluate in situ the sensitivity of mPTP to calcium. In a context of application within clinical protocols, the evaluation of the mPTP calcium sensitivity should contribute to a better understanding of the physiological and physio-pathological mechanisms of adaptation of muscle tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 ;
* Patients referred for a knee ligamentoplasty (DIDT technique) ;
* Patients who signed the non-opposition form after being informed ;
* Patients benefiting from or affiliated to a social security.

Exclusion Criteria:

- Patients under guardianship, curatorship or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for a knee ligamentoplasty
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Determination of the mPTP calcium sensitivity mPTP | day 0
  The goal is to study the feasibility of a new method for the analysis of the calcium sensitivity of mPTP on non-phantomized permeabilized muscle fibers by coupled use of oxygen and fluorimetry techniques. Calcium quantity and time required to open mPTPs in permeabilized muscle fibers will be measured, in the presence or absence of ciclosporin A, observable by total inhibition of mitochondrial respiration (synonymous with release of NADH).

SECONDARY OUTCOMES:
Identification of mPTP opening discrimination factors | Day 0
  Evaluate the possibility of population discrimination by this new method of analysis (i.e. variability by age and duration of functional impotence before intervention of the amount of calcium required to open the mPTP).

CONTACTS AND LOCATIONS:
Overall Officials: Ruddy Richard, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France